CLINICAL TRIAL: NCT07234643
Title: What Matters to You When You Prepare for Surgery and How Does Surgical Preparedness Influence Postoperative Outcome - a Flashmob Study
Brief Title: What Matters to You When You Prepare for Surgery and How Does Surgical Preparedness Influence Postoperative Outcome
Status: Completed | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Horsens Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-16-02-262-25
Record Dates: First submitted 2025-07-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Day Surgery
Keywords: Surgical preparedness; Preoperative worry; Postoperative recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Adult patients undergoing surgery
- Colonoscopy: Adult patients undergoing colonoscopy

SUMMARY:
On the occasion of the international What Matters To You-day 2025 the goal of this Danish, multicenter flashmob study with follow up is to investigate what matters to adult patients when they prepare for surgery or colonoscopy.

Aim

The study has the following aims:

1. To explore and describe what matters to patients when preparing for surgery and to explore how patients prepare before surgery and assess their perceived level of readiness.
2. To examine how the patient's preparation is associated with the quality of their postoperative recovery at home.
3. To examine the associations between Degree of Worry (DOW)/postoperative quality of recovery (QoR-15), and preoperative preparedness/postoperative quality of recovery (QoR-15).

On the day of surgery, patients will be invited to fill out an online questionnaire. At the same time they will be invited to participate in the follow-up on postoperative day 3 (survey link via text message).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical procedures in general anaesthesia, regional anaesthesia, or nerve blocks on June 3th or 6th, 2025, between 7:00 in the morning and 4:00 in the afternoon
* Patients expected to be discharged to their homes the same day.
* ≥18 years old and able to speak and understand Danish.
* For a separate analysis, patients undergoing colonoscopy

Exclusion Criteria:

* Cognitive or psychiatric conditions that impede ability to give informed consent and complete the surveys,
* Non-surgical procedures such as diagnostic endoscopies (with or without biopsy)
* Injection treatments, endovascular treatments or smaller surgical procedures requiring only infiltration analgesia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to ambulatory surgery or colonoscopy in Danish hospitals on June 3rd og June 6th 2025
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Correlation between preoperative preparedness and degree of worry | From enrollment on the day of surgery to postoperative day 3
  The correlation between patients' selfreported preparedness (0 = Not at all prepared, 10 = Very prepared) and the Degree of Worry (0-10 numeric scale, 0 = not all worried and 10 = very worried).

SECONDARY OUTCOMES:
Pre-operative preparation strategies | Baseline
  Multiple choice questions regarding preparation strategies will be asked:
  * Read informational material/watched videos
  * Spoke with healthcare professionals (surgeon, anesthesiologist/nurse anesthetist, others)
  * Spoke with other patients
  * Discussed with family or friends
  * Researched the procedure online
  * Purchased groceries/medications
  * Changed medications
  * Stopped smoking
  * Exercised
  * Avoided infections
  * Arranged for assistance/support from family or friends
  * Planned leave with employer.
Patient preparedness (pre- and postoperatively) | From enrollment on the day of surgery to postoperative day 3
  Patient preparedness (pre- and post-operatively) will be investigated using a numeric rating scale (0 = not at all prepared, 10 = very prepared).
The association between pre-operatively patient preparedness and age | Baseline
  The association between pre-operatively preparedness and age. Patient preparedness will be investigated using a numeric rating scale (0 = Not at all prepared, 10 = Very prepared).
The association between pre-operatively preparedness and gender | Baseline
  The association between pre-operatively preparedness and gender. Patient preparedness will be investigated using a numeric rating scale (0 = not at all prepared, 10 = very prepared).
The association between pre-operatively preparedness and surgical status | Baseline
  The association between pre-operatively preparedness and surgical status will be investigated using a numeric rating scale (0= not at all prepared, 10 = very prepared) and surgical status (elective or acute).
The association between pre-operatively preparedness and living situation | Baseline
  The association between pre-operatively preparedness and living situation (alone/cohabiting). Patient preparedness will be investigated using a numeric rating scale (0 = not at all prepared, 10 = very prepared.
The correlation between pre-operative preparedness and postoperative recovery | From enrollment on the day of surgery to postoperative day 3
  The correlation between pre-operative preparedness shown by a numeric rating scale (0-10) where 0 = "Not a all prepared" and 10 = "Very prepared" and total Quality of Recovery score (QoR-15 score), a 15-item numeric rating scale (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]). A high score indicates a good quality of recovery.
Correlation between preoperative preparedness and degree of Worry | Baseline
  The correlation between pre-operative preparedness shown by a numeric rating scale (0-10) where 0 = "Not a all prepared" and 10 = "Very prepared" and Degree of Worry scale (0-10) where 0 = Not worried at all and 10 = very worried.
What matters when preparing for surgery and was there anything the patient would have known or done differently | From enrollment on the day of surgery to postoperative day 3
  For this outcome a qualitative research approach will be applied. Open-ended responses about What matters when preparing for surgery and was there anything the patient would have known or done differently will be analysed using content analysis focusing on the manifest content
The association between the preparation strategy Read informational material/watched videos and postoperative outcomes | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Read informational material/watched videos and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Spoke with healthcare professionals (surgeon, anesthesiologist/nurse anesthetist, others) and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Spoke with healthcare professionals (surgeon, anesthesiologist/nurse anesthetist, others) and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Spoke with other patients and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Spoke with other patients and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Discussed with family or friends and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Discussed with family or friends and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Researched the procedure online and postoperative outcome | From enrollment of the day of surgery to postoperative day 3
  The association between preparation strategy Researched the procedure online and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy purchased groceries/medications and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy purchased groceries/medications and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Changed medications and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Changed medications and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Stopped smoking and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Stopped smoking and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Exercised and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Exercised and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Avoided infections and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Avoided infections and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Arranged for assistance/support from family or friends and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Arranged for assistance/support from family or friends and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between the preparation strategy Planned leave with employer and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between preparation strategy Planned leave with employer and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The association between other preparation strategies and postoperative outcome | From enrollment on the day of surgery to postoperative day 3
  The association between other preparation strategies and postoperative outcomes: Quality of Recovery - 15 (QoR-15) score and sub scores for Q7 (support from healthcare professionals), Q9 (feel in control), Q14 (anxiety) and Section B of the QoR-15. The scale will be used with each item ranging from 0 to 10 with higher score indicating better QoR. 0 = none of the time [poor] and 10 = all of the time [excellent]).
  The following covariates will be used for the analysis: age, sex, Degree of worry score, surgical status and cohabiting status.
The correlation between Degree of Worry and Quality of Recovery (QoR-15) | From enrollment on the day of surgery to postoperative day 3
  The correlation between the degree of worry shown by the Degree of Worry scale (0-10 numeric scale, 0 = not all worried and 10 = very worried) and QoR-15 scale with each item ranging from 0 to 10 with higher score indicating better QoR (0 = none of the time [poor] and 10 = all of the time [excellent]). The total QoR-15 score and the following individual items will be used:Q7 (support from healthcare professionals), Q9 (feel in control), Q10 (feeling of well-being), Q14 (anxiety) as well as section B.

OTHER OUTCOMES:
Quality of Recovery score (QoR-15) | On postoperative day 3
  Quality of Recovery score (QoR-15), a 15-item numeric rating scale (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]). A high score indicates a good quality of recovery. Results will be summarized using percentages, means with standard deviations, or medians with interquartile ranges (IQR) for the entire population.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Nielsen, PhD, Study Chair — Gødstrup Hospital
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Gødstrup Hospital, Herning
  - Horsens Hospital, Horsens

IPD SHARING:
Plan to Share IPD: Yes
Demographics:
  Age, gender, status of procedure (emergency/planned), surgical specialty, hospital, living situation (alone/cohabiting), phone number for survey distribution via text message.
  Preparation-related questions:
  * What matters to you when preparing for surgery? Open ended response
  * How have you prepared for the surgery? Response format: Multiple-choice checkboxes
  * How worried are you about the first few post-operative days? Response format: Degree of Worry, 0-10 numeric rating scale
  Quality of Recovery score (QoR-15)
  Retrospective preparation assessment:
  * Looking back, how well-prepared were you for surgery? Response format: 0-10 numeric rating scale
  * Was there anything you wish you had known or done? Response format: Multiple choice categories + option for open ended response
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date: June 3 2025 End date: January 2026
Access Criteria: Data will be collected through the REDCap database. Collaborators in the steering group will be granted access to all data in the REDCap database.
  Collaborators who enroll patients to the study from various Danish locations will be provided with data from their specific location/site. They will not be provided with access to REDCap but will receive data in a data file.